CLINICAL TRIAL: NCT01018836
Title: A Phase I Trial of Riluzole in Combination With Radiation Therapy in Patients Undergoing Whole Brain Radiation Therapy for Brain Metastasis
Brief Title: Riluzole and Whole-Brain Radiation Therapy in Treating Patients With Brain Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050808; CDR0000660044 (Other: NIH); P30CA072720 (NIH)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riluzole; Radiation Therapy (Experimental)
  Interventions: Drug: riluzole; Radiation: whole-brain radiation therapy

INTERVENTIONS:
Drug: riluzole — The first dose of Riluzole will be day 0 of study enrollment. WBRT must begin within 48 hours of the initiation of Riluzole therapy. At the completion of radiation, Riluzole should be discontinued and steroids should be tapered over the course of 1-3 weeks, at the discretion of the treating physicians.
Radiation: whole-brain radiation therapy — Standard whole brain irradiation will be carried out at 250 cGy per day fractions times 15 to a total dose of 3750 cGy using a standard opposed lateral helmet field with the inferior border inclusive of C1.

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. Drugs, such as riluzole, may make tumor cells more sensitive to radiation therapy. Giving riluzole together with whole-brain radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of riluzole when given together with whole-brain radiation therapy in treating patients with brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of riluzole that can be administered concurrently with standard whole-brain radiotherapy (WBRT) in patients with multiple brain metastases.

Secondary

* To determine the long-term toxicity of riluzole when administered with WBRT.
* To assess neurocognitive function before and after treatment with riluzole and WBRT.
* To determine the MRI response of brain metastasis after treatment with riluzole and WBRT.
* To compare survival of patients treated with riluzole and WBRT to published historical data for patients with brain metastases.
* To evaluate the response of brain metastasis to riluzole and WBRT as a function of the expression of glutamate receptors on the primary tumor specimen.

OUTLINE: This is a dose-escalation study of riluzole.

Patients receive oral riluzole twice daily beginning on day 0. Beginning within 2 days after the initiation of riluzole, patients undergo whole-brain radiotherapy for 15 fractions.

Patients undergo neurocognitive and quality-of-life assessments at baseline, at 5 weeks, and at 3 months.

Tumor tissue samples are collected for laboratory biomarker studies.

After completion of study treatment, patients are followed up at 6 weeks, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor
* Has ≥ 2 brain metastases as demonstrated by baseline MRI

  * Patients with only 1 metastasis are eligible provided the metastasis is too large for radiosurgery and not amenable to surgical resection
* Not being considered for surgical resection
* Eligible to undergo whole-brain radiotherapy (WBRT)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,000/μL
* Platelet count ≥ 50,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 1.5 times ULN
* INR ≤ 1.5 times ULN
* Sodium normal
* Thyroid-stimulating hormone normal
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for ≥ 6 months after completion of study treatment
* No headaches, disequilibrium, vertigo, or dizziness
* No known history of hepatitis B or C
* No concurrent serious systemic disorder (including active infection) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* No history of allergic reactions attributed to riluzole

PRIOR CONCURRENT THERAPY:

* No prior WBRT
* At least 2 weeks since prior systemic chemotherapy
* No systemic chemotherapy during and for ≥ 3 weeks after completion of WBRT
* Radiosurgical boosts to ≤ 3 metastases allowed, based on the discretion of the treating radiation oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of riluzole | 2.5 years

SECONDARY OUTCOMES:
Long-term toxicity of riluzole | .25 years
Neurocognitive function before and after treatment | 2.5 years
MRI response of brain metastasis after treatment | 2.5 years
Survival | 2.5 years
Response of brain metastasis to treatment as a function of the expression of glutamate receptors | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Haffty, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States